CLINICAL TRIAL: NCT04267965
Title: Changes of Pulmonary Function, Voice and Swallowing Symptoms After Total Parathyroidectomy for Secondary Hyperparathyroidism in the Presence of Intact Recurrent Laryngeal Nerve
Brief Title: Pulmonary Function, Voice and Swallowing Symptoms After Parathyroidectomy
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chou Fong-Fu, Consultant professor, Chang Gung Memorial Hospital
Other Study IDs: 201601901B0
Record Dates: First submitted 2020-01-22; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Secondary Hyperparathyroidism Due to Renal Causes
Keywords: Voice impairment; airway invasion; respiratory function
MeSH Terms: conditions — Dysphonia; Respiratory Aspiration | interventions — Parathyroidectomy; Transplantation, Autologous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients who have been successfully operated on with total parathyroidectomy for symptomatic secondary hyperparathyroidism and their PTH levels are below 72 pg/dL within one week after surgery.
  Interventions: Procedure: parathyroidectomy plus bilateral thymectomy and autotransplantation
- Group B: Patients who have had regular dialysis and their iPTH levels are around 500 pg/dL

INTERVENTIONS:
Procedure: parathyroidectomy plus bilateral thymectomy and autotransplantation — Patients should receive total parathyroidectomy plus bilateral thymectomy and autotransplantation
  Groups: Group A

SUMMARY:
In this study, investigators measure patient's voice frequency, swallowing function, and O2 desaturation of the 6 mins walking test before surgery and 4 months after surgery, to find the increase of voice frequency, and swallowing function and the decrease of O2 desaturation.

DETAILED DESCRIPTION:
This was a prospective case-control study. From July 2017 to Dec. 2018, investigators recruited 38 patients, who had undergone a successful operation of total parathyroidectomy and bilateral thymectomy (TPxBT) plus autotransplantation for symptomatic secondary hyperparathyroidism as the study group. In the same period 4 patients who had a surgical failure were excluded from the study. Indications for surgery were patients who had undergone long-term regular hemodialysis or continuous ambulatory peritoneal dialysis (CAPD), with serum levels of Ca > 10.1 mg/dL, P > 5.5 mg/dL, alkaline phosphatase (Alk-ptase) > 94 U/L and intact parathyroid hormone(iPTH) > 800 pg/mL and with symptoms and signs such as skin itching, bone pain, general weakness, insomnia and T-score of bone mineral density (BMD) (the lowest T-score of lumbar spine 1-4, global femur, femoral neck, radial 1/3, and global radius) < -2.5. During surgery, Total parathyroidectomy and bilateral thymectomy was performed plus autotranplantation of 100 mg of hyperplastic parathyroid tissue to the subcutaneous tissue of the forearm without harboring an arteriovenous fistula.

Ten patients with regular hemodialysis who had developed mild secondary hyperparathyroidism (iPTH around 500 pg/mL) but did not undergo parathyroidectomy were recruited as the control group.

Investigators recorded patients' age, symptoms, gender, body mass index (BMI) and measured serum levels of Ca, P, Alk-ptase and iPTH, and BMD (T-score). The Investigators also recorded patients' voice quality, airway invasion during swallowing and pulmonary functions before surgery and 4 months after surgery to find the changes after surgery. In the control group, investigators recorded and measured these items at baseline and 4 months later.

At 1 week after surgery, serum Ca, P, Alk-ptase and iPTH levels were measured again to make sure that the operation was successful. A successful operation was defined as iPTH levels < 72 pg/mL within 1 week after surgery. Four patients were excluded from this study with a surgical failure in the same period.

The perceptual evaluation of voice quality such as speech impairment and speech quality by means of multidimensional clinical measurements based on auditory methods with grade, hoarseness, roughness, breathiness, asthenia, and strain (GRBAS) on a scale (0-3) (normal-high degree) were performed by the ear, nose, and throat specialist (Dr. Lai, C.C.). Voice handicap index (VHI-10) (>11, abnormal) and eating assessment tool (EAT-10) (≥ 3, abnormal) were evaluated by patients themselves.

Acoustic and aerodynamic measurements were applied to recordings of each subject producing sustained vowel productions in a soundproof room. Acoustic variables including jitter (Jitt), shimmer (ShdB), noise-to-harmonic ratio (NHR), fundamental frequency (Fo), and high pitch were measured using computerized speech laboratory (Core Model SCL # 4300B, KayPENTAX Elementries, Lincoln park, NJ).

The maximal phonation time and s/z ratio were measured with circumferentially vented pneumotachography mask and differential transducers of the Aerophone system (Aerophone II, Model 6800, KayPENTAX Elementrics). Vocal cord mobility, vocal cord closure (complete or incomplete), airway invasion during swallowing were inspected with fiber-optic endoscopy to show premature spillage, penetration-aspiration scale levels (1-8) (no entry of material into the larynx or trachea-material enter the airway passes below vocal folds and no effort is made to eject) (>1, abnormal). The Yale pharyngeal residue severity rating scale for vallecula (0-4) (non-trace-mild-moderate-severe) and pyriform sinus (0-4) were also performed by the ENT specialist.

The specialist of chest medicine (Dr. Chang, H.C.) performed pulmonary function tests including forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), bronchodilator test (BDT) (a positive response to BDT defined by the American Thoracic Society as an increase in FEV1 or FVC ≥ 12% and 200 ml), total lung capacity (TLC), and alveolar volume (VA) using MasterScope (Jaeger, VIASYS healthcare GmbH, Höchberg, Germany), and diffusion capacity of the lung for carbon monoxide (DLCO) using Vmax Autobox (SensorMedics, a subsidiary of VIASYS healthcare, California, USA). The 6 minutes walking test (6MWT) was also performed to evaluate distance (meter) and O2 desaturation (differences of O2 saturation between pre- and post-tests) (defined as positive if O2 desaturation ≧ 4%).

ELIGIBILITY:
Inclusion Criteria:

1. age over 20 years
2. chronic renal failure with regular dialysis
3. iPTH> 800pg/mL, Ca > 10.1 mg/dL, and P > 5.5 mg/dL
4. symptoms of bone pain, skin itching, general weakness, insomnia and osteoporosis (T score< -2.5)

Exclusion Criteria:

1. pregnancy women
2. patients after kidney transplantation
3. a failure in surgery

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We included patients who had symptomatic secondary hyperparathyroidism and were successfully operated during the two years period (Aug 1 2017 - July 31 2019).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Successful surgery is defined as iPTH levels less than 72 pg/dL within one week after surgery | one week after surgery
  After successful surgery, patients were recruited in the study, and we excluded patients with a surgical failure.
Voice impairment(GRBAS) | 4 months after surgery
  speech impairment and speech quality were evaluated with GRBAS on a scale (0-3), VHI-10 (>11, abnormal) and (EAT-10) (≥ 3, abnormal) .
  *GRBAS (grade, roughness, breathiness, asthenia, strain) scale grades hoarseness, roughness, breathiness, aesthenia (weakness), and strain on a scale of 0-3 0 = normal, 1 = mild degree, 2 = moderate degree, and 3 = high degree
Voice impairment(VH1-10) | 4 months after surgery
  speech impairment and speech quality were evaluated with voice handicap index (VHI-10) (>11, abnormal) 0-4 Rating Scale 0 = Normal
  1. = Almost Normal
  2. = Sometimes
  3. = Abnormal
  4. = Always
Voice impairment(EAT-10) | 4 months after surgery
  speech impairment and speech quality were evaluated with EAT-10 (≥ 3, abnormal) .
  *eating assessment tool (EAT-10) 0 - 4 Rating Scale 0 = No problem
  1. = Mild Problem
  2. = Mild to moderate
  3. = Moderate problem
  4. = Severe problem
Acoustic voice analysis | 4 months after surgery
  mean frequency (F0, Hz); Noise-to-Harmonic Ratio (NHR), jitter(%), and shimmer (%)
Vocal cord examination | 4 months later
  The maximal phonation time (sec) and s/z ratio were measured with circumferentially vented pneumotachography mask and differential transducers of the Aerophone system .
Fiber optic endoscopic evaluation of swallowing (FEES) | 4 months later.
  Vocal cord mobility, vocal cord closure (complete or incomplete), airway invasion during swallowing were inspected with fiber-optic endoscopy to show premature spillage, penetration-aspiration scale levels . The Yale pharyngeal residue severity rating scale for vallecula and pyriform sinus (0-4) (non-trace-mild-moderate-severe) and pyriform sinus (0-4) were also performed.
Pulmonary function test | 4 months later
  Forced vital capacity (FVC) (L), forced expiratory volume in 1 second (FEV1), bronchodilator test (BDT) (a positive response to BDT defined by the American Thoracic Society as an increase in FEV1 or FVC ≥ 12% and 200 ml), total lung capacity (TLC) (L), and alveolar volume (VA) using MasterScope (Jaeger, VIASYS healthcare GmbH, Höchberg, Germany), and diffusion capacity of the lung for carbon monoxide (DLCO) (%) using Vmax Autobox (SensorMedics, a subsidiary of VIASYS healthcare, California, USA).
6MWT were performed. | 4 months later
  The 6 minutes walking test (6MWT) was also performed to evaluate distance (meter) and O2 desaturation (differences of O2 saturation between pre- and post-tests) (defined as positive if O2 desaturation ≧ 4%).

CONTACTS AND LOCATIONS:
Overall Officials: Chang Huang-Chih, MD, Study Director — Co-host; Chen Jib-Bor, MD, Study Director — Co-host; Lai Chi-Chih, MD, Study Director — Co-host
Locations (1):
- Fong-Fu Chou, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Okada M, Tominaga Y, Yamamoto T, Hiramitsu T, Narumi S, Watarai Y. Location Frequency of Missed Parathyroid Glands After Parathyroidectomy in Patients with Persistent or Recurrent Secondary Hyperparathyroidism. World J Surg. 2016 Mar;40(3):595-9. doi: 10.1007/s00268-015-3312-1. PMID 26563219
- [Result] Wood JM, Athanasiadis T, Allen J. Laryngitis. BMJ. 2014 Oct 9;349:g5827. doi: 10.1136/bmj.g5827. No abstract available. PMID 25300640
- [Result] Arffa RE, Krishna P, Gartner-Schmidt J, Rosen CA. Normative values for the Voice Handicap Index-10. J Voice. 2012 Jul;26(4):462-5. doi: 10.1016/j.jvoice.2011.04.006. Epub 2011 Aug 4. PMID 21816570
- [Result] Belafsky PC, Mouadeb DA, Rees CJ, Pryor JC, Postma GN, Allen J, Leonard RJ. Validity and reliability of the Eating Assessment Tool (EAT-10). Ann Otol Rhinol Laryngol. 2008 Dec;117(12):919-24. doi: 10.1177/000348940811701210. PMID 19140539
- [Result] Eckel FC, Boone DR. The S/Z ratio as an indicator of laryngeal pathology. J Speech Hear Disord. 1981 May;46(2):147-9. doi: 10.1044/jshd.4602.147. PMID 7253591
- [Result] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Result] Neubauer PD, Rademaker AW, Leder SB. The Yale Pharyngeal Residue Severity Rating Scale: An Anatomically Defined and Image-Based Tool. Dysphagia. 2015 Oct;30(5):521-8. doi: 10.1007/s00455-015-9631-4. Epub 2015 Jun 7. PMID 26050238
- [Result] Richter DC, Joubert JR, Nell H, Schuurmans MM, Irusen EM. Diagnostic value of post-bronchodilator pulmonary function testing to distinguish between stable, moderate to severe COPD and asthma. Int J Chron Obstruct Pulmon Dis. 2008;3(4):693-9. doi: 10.2147/copd.s948. PMID 19281083
- [Result] Single breath carbon monoxide diffusing capacity (transfer factor). Recommendations for a standard technique. Statement of the American Thoracic Society. Am Rev Respir Dis. 1987 Nov;136(5):1299-307. doi: 10.1164/ajrccm/136.5.1299. No abstract available. PMID 3674590
- [Result] Waatevik M, Johannessen A, Gomez Real F, Aanerud M, Hardie JA, Bakke PS, Lind Eagan TM. Oxygen desaturation in 6-min walk test is a risk factor for adverse outcomes in COPD. Eur Respir J. 2016 Jul;48(1):82-91. doi: 10.1183/13993003.00975-2015. Epub 2016 Apr 13. PMID 27076586